CLINICAL TRIAL: NCT01057602
Title: Further Validation of the Memory Orientation Screening Test (MOST): A 5-minute Screening Test for Dementia in Primary Care Practice
Brief Title: Further Validation of the Memory Orientation Screening Test (MOST):A 5-minute Screening Test for Dementia in Primary Care Practice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clionsky, Mitchell, Ph.D., ABPP(CN) (Individual)
Responsible Party: Mitchell Clionsky, Ph.D., Clionsky Neuro Systems, LLC
Other Study IDs: SP2008-004
Record Dates: First submitted 2010-01-23; First posted 2010-01-27 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-01

CONDITIONS: Dementia
Keywords: Dementia; Screening Tests; Cognition; Memory; MOST
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Normal community dwelling elders: Individuals age 65 and older who live in the community

SUMMARY:
The purpose of this study is to apply a recently developed screening test for dementia, the Memory Orientation Screening Test (MOST) to two additional groups. Group one is composed of 150 elders who do not have dementia and are residing in the community so that we can determine what is a "normal" MOST score. These subjects will also be individually administered a one-hour battery composed of other commonly used tests of memory and information processing. Group two is composed of 150 elders who are administered the MOST by a nurse as part of their regular visit to the primary care doctor's office, and their scores will be compared against a rating of their cognitive ability made independently by the doctor or another nurse. Their scores will also be compared with a list of their medical problems and medications. Our hypothesis for the first group is that the MOST scores will be higher in the normal group than in the previous clinical groups and that MOST scores will correlate significantly with other neurocognitive tests. Our hypothesis for the second group is that the MOST can be administered quickly and easily by briefly trained nurses, that it will compare highly with doctor opinions, and that patients with known medical conditions related to dementia, such as hypertension or diabetes, will have lower MOST scores than patients in better health.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older

Exclusion Criteria:

* Younger than 65,
* diagnosed with dementia,
* blind,
* non-English speaking

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community sample and primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Memory Orientation Screening Test score | Day 1

SECONDARY OUTCOMES:
Other neuropsychological test scores and doctor ratings | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell I Clionsky, Ph.D., Principal Investigator — Clionsky Neuro Systems
Locations (1):
- Clionsky Neuro Systems, LLC, Springfield, Massachusetts, United States